CLINICAL TRIAL: NCT05667064
Title: Specific Use-results Study of IMJUDO Intravenous Infusion 25 mg, 300 mg / IMFINZI Intravenous Infusion 120 mg, 500 mg All Patient Investigation in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Imfinzi/Imjudo uHCC Japan PMS _ Japan Post-Marketing Surveillance (PMS) Study
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419CC00026
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Unresectable Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
This investigation will be conducted to collect information of safety in patients with unresectable hepatocellular carcinoma (HCC) treated with the combination therapy of IMJUDO 25 mg, 300 mg and IMFINZI Intravenous Infusion 120 mg, 500 mg or with IMFINZI monotherapy under actual use in the post-marketing setting.

DETAILED DESCRIPTION:
This investigation will be conducted to collect information of safety in patients with unresectable hepatocellular carcinoma (HCC) treated with the combination therapy of IMJUDO 25 mg, 300 mg and IMFINZI Intravenous Infusion 120 mg, 500 mg or with IMFINZI monotherapy under actual use in the post-marketing setting.

The investigation will be conducted as one of the additional pharmacovigilance activities in the Japan Risk Management Plan of IMJUDO and IMFINZI in compliance with the Ministerial Ordinance on Good Post-marketing Study Practice (GPSP Ordinance) and for the purpose of application for reexamination under Article 14-4 of the Act on Securing Quality, Efficacy and Safety of Products Including Pharmaceuticals and Medical Devices.

ELIGIBILITY:
Inclusion Criteria:

All patients who receive IMJUDO and IMFINZI combination therapy or IMFINZI monotherapy for their unresectable HCC.

-

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unresectable HCC
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of ADRs | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (47):
- Japan (47):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home